CLINICAL TRIAL: NCT05460767
Title: A Phase Ia/Ib Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of IBI363 in Subjects With Advanced Solid Tumors or Lymphoma
Brief Title: Safety, Tolerability and Preliminary Efficacy of IBI363 in Subjects With Advanced Solid Tumors or Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363A102
Record Dates: First submitted 2022-07-05; First posted 2022-07-15 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumors or Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI363 (Experimental): Single arm
  Interventions: Biological: IBI363

INTERVENTIONS:
Biological: IBI363 — a mutated IL-2 cytokine fused to an anti-PD-1 antibody to combine IL-2 pathway stimulation with checkpoint blockade.

SUMMARY:
This study is an open-label, multicenter, phase Ia/Ib study. The study will evaluate the safety, tolerability and preliminary efficacy of IBI363 in subjects with advanced, relapsed or metastatic solid tumors or lymphoma, determine the maximum tolerated dose (MTD) or maximum administered dose (MAD), and thus determine the recommended phase 2 dose (RP2D).

DETAILED DESCRIPTION:
This study is an open-label, multicenter, phase Ia/Ib study. The study will evaluate the safety, tolerability and preliminary efficacy of IBI363 in subjects with advanced, relapsed or metastatic solid tumors or lymphoma, determine the maximum tolerated dose (MTD) or maximum administered dose (MAD), and thus determine the recommended phase 2 dose (RP2D). The phase Ia part consists of the dose escalation and PD marker exploration part. The phase Ib part consists of the dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ≥ 18 years
2. Histologically or cytologically confirmed, unresectable locally advanced or metastatic solid tumors or lymphomas
3. Subjects who progressed or are intolerant to existing standard therapy or subjects without standard therapy Note: Subjects may have received and failed prior therapy with a PD-1/PD-L1 inhibitor and be considered eligible for this trial.
4. Subjects with at least one measurable lesion according to RECIST v1.1 for solid tumor or Lugano 2014 for lymphoma
5. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
6. Expected survival time ≥ 3 months.

Exclusion Criteria:

1. Subjects with history of or known active seizure disorder, brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
2. Subjects with active thrombosis, or a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within 4 weeks prior to first administration of study drug unless adequately treated and considered by the Investigator to be stable.
3. Active uncontrolled bleeding or a known bleeding diathesis.
4. Subjects with massive pleural effusion or massive ascites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of dose-limiting toxicity (DLT) | 21 days during the first 3-week cycle
  Incidence of dose-limiting toxicity (DLT) events
incidence of adverse enents (AE), serious adverse events (SAEs), treatment-emergent AEs (TEAEs) and immune-related AEs (irAEs) | up to 90 days after the last administration
  AE is defined as an unexpected medical problem that happens during treatment with a drug or other therapy. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is an important medical event that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before. A TEAE will be defined as any new AE that begins, or any pre-existing condition that worsens in severity, after at least 1 dose of study treatment has been administered. irAEs will be assessed.
Number of participants with abnormality in vital signs | up to 90 days after the last administration
  Blood pressure, pulse, respiratory rate, and temperature will be assessed.
Number of participants with abnormality in hematology parameters | up to 90 days after the last administration
  Blood samples will be collected to evaluate hemoglobin, white blood cell (WBC) count, platelets and coagulation factors including international normalized ratio (INR), activated partial thromboplastin time (aPTT) and prothrombin time (PT)
Number of participants with abnormality in clinical chemistry parameters | up to 90 days after the last administration
  Blood samples will be collected to evaluate sodium, potassium, calcium, magnesium, chloride, glucose, creatinine, urea or blood urea nitrogen (BUN), bicarbonate, amylase, bilirubin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total protein, albumin, lactate dehydrogenase and lipase.
Number of participants with abnormality in routine urinalysis parameters | up to 90 days after the last administration
  Urine samples will be collected to evaluate specific gravity, leucocyte esterase, nitrite, blood, bilirubin, protein, glucose, ketones and urobilinogen.
Number of participants with abnormality in ECG parameters | up to 90 days after the last administration
  12-lead ECG will be obtained using an ECG machine. Participants will be in supine or a semi-recumbent position (about 30 degrees of elevation) and rested for approximately 2 minutes before ECGs are recorded.

SECONDARY OUTCOMES:
maximum concentration (Cmax) | Up to 2 years
  PK parameters to be evaluated for IBI363 including maximum concentration (Cmax) will be determined when appropriate.
area under the curve (AUC) | Up to 2 years
  PK parameters to be evaluated for IBI363 including area under the curve (AUC) will be determined when appropriate.
clearance (CL) | Up to 2 years
  PK parameters to be evaluated for IBI363 including clearance (CL) will be determined when appropriate.
half-life (t1/2) of IBI363 | Up to 2 years
  PK parameters to be evaluated for IBI363 including half-life (t1/2) will be determined when appropriate.
volume of distribution (V) | Up to 2 years
  PK parameters to be evaluated for IBI363 including volume of distribution (V) will be determined when appropriate.
Objective response rate (ORR) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
time to response (TTR) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
duration of response (DoR) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
disease control rate (DCR) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
progression-free survival (PFS) | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
6-month and 1-year PFS rate | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
Overall survival (OS) | through study completion, an average of 1 year
  To evaluate the preliminary antitumor activity of IBI363
6-month and 1-year OS rate | Up to 2 years
  To evaluate the preliminary antitumor activity of IBI363
The incidence of ADA and NAb of IBI363 | Up to 2 years
  Each subject will be tested for anti-drug (IBI363) antibody (ADA), and ADA-positive serum samples will continue to be tested for neutralizing antibodies (NAb).

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China